CLINICAL TRIAL: NCT01697618
Title: A Randomised, Double-blind, Single Centre, Two-way Cross-over Trial Comparing the Pharmacokinetics, Pharmacodynamics and Safety of the Biphasic Insulin Aspart 30 and Insulin Mixtard 30/70 After Multiple Dosing With a Twice Daily Dose Regimen in Type 2 Diabetic Patients
Brief Title: Pharmacokinetics, Pharmacodynamics and Safety of Biphasic Insulin Aspart 30 in Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ANA/DCD/046
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic human insulin 30
- BHI 30 (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic human insulin 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Injected subcutaneously (s.c., under the skin) before breakfast and dinner, dosage adjusted throughout the trial according to individual needs
Drug: biphasic human insulin 30 — Injected subcutaneously (s.c., under the skin) before breakfast and dinner, dosage adjusted throughout the trial according to individual needs

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate pharmacokinetics, pharmacodynamics and safety of biphasic insulin aspart 30 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months
* Treated with a combination of soluble/protracted human insulin in the ratio of 30/70 in a twice-daily regimen for at least 6 months
* BMI (body mass index) below 39 kg/m^2
* HbA1c (glycosylated haemoglobin) below 12%

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1997-04; Primary Completion 1998-11 (Actual); Study Completion 1998-11 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin curve

SECONDARY OUTCOMES:
Overall shape of the 24 hour serum insulin profile
Cmax (maximum plasma concentration)
tmax (time to reach maximum)
Area under the curve following each injections derived from 24 hours serum insulin profiles
Overall shape of the 24 hour serum glucose profile
Serum glucose excursions (EXC)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (2):
- Novo Nordisk Investigational Site, Alphen aan den Rijn, Netherlands
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- [Result] McSorley PT, Bell PM, Jacobsen LV, Kristensen A, Lindholm A. Twice-daily biphasic insulin aspart 30 versus biphasic human insulin 30: a double-blind crossover study in adults with type 2 diabetes mellitus. Clin Ther. 2002 Apr;24(4):530-9. doi: 10.1016/s0149-2918(02)85129-3. PMID 12017398
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com